CLINICAL TRIAL: NCT07272005
Title: Improving Control of Intermittent Exotropia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Responsible Party: Principal Investigator, Eileen Birch, Director, Pediatric Vision Laboratory, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03 IXT2 2026
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Dichoptic Videos (Experimental): dichoptic videos streamed at home 1 hour per day, 5 days per week
  Interventions: Other: dichoptic videos
- Group 2: Standard Videos (Sham Comparator): standard videos streamed at home 1 hour per day, 5 days per week
  Interventions: Other: standard videos

INTERVENTIONS:
Other: dichoptic videos — custom designed dichoptic videos
  Arms: Group 1: Dichoptic Videos
Other: standard videos — standard videos
  Arms: Group 2: Standard Videos

SUMMARY:
To determine whether use of dichoptic movies for 8 weeks may be helpful in improving control alignment in children with intermittent exotropia (IXT), thus allowing IXT to be managed non-surgically

DETAILED DESCRIPTION:
Intermittent exotropia (IXT) is the most common form of strabismus, characterized by an outward deviation of the eyes that is primarily manifest during distance fixation and can intermittently be controlled by fusional mechanisms. Less than 30% of children have good long-term outcomes following treatment for spontaneously manifest IXT with current non-surgical treatments (prism therapy, over-minus lenses, or vision therapy). The limited efficacy of current non-surgical treatments for IXT is thought to arise from underlying sensory deficits, particularly interocular suppression, which compromises binocular function. This underscores the need for sensory-directed interventions aimed at reducing suppression and thereby enhancing the potential for stable binocular outcomes.

In this study, children will be randomized to watch engaging videos streamed at home that are either dichoptic or standard (control) format. The aim is to determine whether the dichoptic format will decrease suppression and improve control of eye alignment . In previous research, use of dichoptic games and movies by children with amblyopia has shown to reduce suppression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IXT or XT at Distance & IXT or XP at near (Basic or Pseudo Divergence Excess subtype of IXT)
* No surgery planned for 6 months

Exclusion Criteria:

* Prior eye muscle surgery
* Prior binocular treatment or vision therapy
* Amblyopia
* Neurological conditions, seizure disorders, vestibular abnormalities, or frequent headache
* Other eye conditions (refractive error OK)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in control of intermittent exotropia | 8 weeks
  change percent time alignment is present at 8 weeks vs at baseline

SECONDARY OUTCOMES:
Improvement in control of intermittent exotropia | 4 weeks
  change percent time alignment is present at 4 weeks vs at baseline
Improvement in control of intermittent exotropia | 12 weeks off-treatment
  change percent time alignment is present at 12 weeks off-treatment weeks vs at baseline
Change in suppression | 4 weeks
  change in HATT test score at 4 weeks vs at baseline
Change in suppression | 8 weeks
  change in HATT test score at 8 weeks vs at baseline
Change in suppression | 12 weeks off-treatment
  change in HATT test score at 12 weeks off-treatment vs at baseline
Change in distance stereoacuity | 4 weeks
  change in Distance Randot test score at 4 weeks vs at baseline
Change in distance stereoacuity | 8 weeks
  change in Distance Randot test score at 8 weeks vs at baseline
Change in distance stereoacuity | 12 weeks off-treatment
  change in Distance Randot test score at 12 weeks off-treatment vs at baseline
Change in quality of life | 8 weeks
  Change in IXTQ questionnaire (Rasch-scored on a 0-100 scale) at 8 weeks vs at baseline
Change in quality of life | 12 weeks off-treatment
  Change in IXTQ questionnaire (Rasch-scored on a 0-100 scale) ay 12 weeks off-treatment vs at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eileen E Birch, Principal Investigator — Retina Foundation of the Southwest

IPD SHARING:
Plan to Share IPD: No